CLINICAL TRIAL: NCT03141931
Title: The Effects of Dietary Supplementation With a Combination of Flaxseed Oil, Borage Oil and Fish Oil Omega-3 Fatty Acids on Ocular Comfort Including Symptoms of Dry Eye
Brief Title: The Effects of Dietary Supplementation With Omega-3 Fatty Acids on Symptoms of Dry Eye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of New South Wales (Other)
Responsible Party: Principal Investigator, Jacqueline Tan-Showyin, Senior Research Fellow, The University of New South Wales
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SOVS2016-045
Record Dates: First submitted 2017-02-06; First posted 2017-05-05 (Actual); Results first posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-05

CONDITIONS: Dry Eye
Keywords: Nutraceutical supplement
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplement (Experimental): Combination of flaxseed oil, borage oil and fish oil omega-3 fatty acids
  Interventions: Dietary Supplement: Supplement
- Placebo (Placebo Comparator): Polyethylene glycol, Oleic acid, Propylene glycol
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Supplement — Concentrated Omega-3 Triglycerides-fish 332 mg Equiv. Eicosapentaenoic Acid (EPA) 134 mg Equiv. Docosahexaenoic Acid (DHA) 66.8 mg Flax Seed Oil (Linseed Oil) 334 mg Equiv. Oleic acid 58.5 mg Equiv. Linoleic acid 58.5 mg Equiv. Linolenic acid 192 mg Borago officinalis seed oil fixed (Borage) 434 mg Equiv. gamma-Linolenic acid 95.5 mg
  Arms: Supplement
Dietary Supplement: Placebo — polyethylene glycol (500mg), oleic acid (659mg) and propylene glycol (115mg)
  Arms: Placebo

SUMMARY:
The aim of this study is to compare ocular symptoms and signs when the test nutraceutical formulation (combination of flaxseed oil, borage oil and fish oil omega-3 fatty acids) is consumed daily over a 3 month period, with a control capsule that contains polyethylene glycol (PEG), oleic acid and propylene glycol, which are found in many pharmaceutical products and are generally considered to be biologically inert and safe. There is good evidence that the consumption of oily fish has a protective effect against dry eye, and other studies have provided evidence of the beneficial effect of supplementation with omega-3 essential fatty acids in the treatment of dry eye disease. However, there have been limited well designed clinical trials investigating the potential for nutraceutical dietary supplementation to impact ocular comfort. To date, no controlled, randomised clinical trials have been conducted to evaluate the test nutraceutical formulation. Therefore, the purpose of this study is to conduct a randomized, placebo-controlled, double-masked study to investigate the effects of dietary supplementation with a combination of flaxseed oil, borage oil and fish oil omega-3 fatty acids on ocular comfort including signs and symptoms of dry eye.

DETAILED DESCRIPTION:
This study will be a prospective, randomised, placebo-controlled, double masked study conducted over a 3-month period. One hundred and thirty-eight (138) participants who meet the inclusion / exclusion criteria and give informed consent will be randomised to either the test capsules containing a combination of flaxseed oil, borage oil and fish oil omega-3 fatty acids or placebo capsules, identical in appearance, containing polyethylene glycol, oleic acid and propylene glycol (found in many pharmaceutical products and considered to be biologically inert and safe) to be taken by mouth three times daily for 40 days, and then twice daily thereafter for approximately 50 days. Every effort will be made to stratify enrolment by disease severity to ensure participants with mild, moderate and severe dry eye are represented in the study population. Stratification will be in a 2:2:1 fashion i.e. OSDI score >12 (55 participants), OSDI score >20 (55 participants) and OSDI score >45 (28 participants). Participants will be stratified according to dry eye severity prior to randomisation. There will be a total of 3 scheduled study visits over a period of approximately 3 months - Day 1, 1 month and 3 months. Ocular comfort and symptoms of dry eye will be assessed via questionnaires. The tear film and ocular surface will be assessed using specialised instruments including the slit lamp biomicroscope, Lipiview Ocular Surface Interferometer, Vapometer and Oculus Keratograph 5M, and stains. Safety will be assessed through measurement of vision, ocular redness and evaluation of the ocular surface using the slit lamp biomicroscope. Those participants who meet the eligibility criteria will be randomly allocated to either the test or control capsules. An adequate supply of capsules will be dispensed to last until the next Participants will be instructed to ingest one capsule three times daily with meals for 40 days, and then two times daily until their final 3 month study visit.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and comprehend English and give informed consent as demonstrated by signing a record of informed consent;
* Be at least 18 years old;
* Have symptoms of ocular discomfort as measured with the Ocular Surface Disease Index (OSDI) score of >12 at the Baseline visit;
* Willing to comply with the dosage and study visit schedule as directed by the investigator;
* No contact lens wear in the last 30 days and willing to refrain from contact lens wear for the duration of the study;
* No planned changes to diet and willing not to substantially alter their usual diet for the duration of the study, including their typical intake of fish;
* Willingness to notify the study investigator if instructed to alter their diet by health/medical practitioner;
* Willing to continue using any artificial tear supplements at the same frequency throughout the study, as used prior to the study
* Have health and ocular health findings which would not prevent the participant from safely ingesting dietary supplementation with combination omega oils

Exclusion Criteria:

* Any systemic disease that would preclude participants from safely ingesting dietary supplementation with combination omega oils;
* Self-reported allergy/sensitivity to any of the study product ingredients;
* Use of any polyunsaturated fatty acid-containing dietary supplements (such as fish oil, evening primrose oil, linseed oil) up to 12 weeks prior to the start of the study;
* Use of any of the following medications (including steroids) up to 12 weeks prior to start of the study or during the course of the study:

  * Ocular medication, category S3 and above;
  * Any systemic or topical medications that will affect ocular physiology e.g. anti-acne medications such as Roaccutane and corticosteroid or immunosuppressant medications such as Hydrocortisone, Prednisolone and antihistamine medications such as Claritine;
* Any systemic disease that may affect ocular health e.g. Graves disease, and auto-immune diseases such as ankolysing spondylitis, multiple sclerosis and systemic lupus erythematosis;
* Epilepsy or history of migraines exacerbated by flashing, strobe-like lights;
* Eye surgery within 6 months immediately prior to enrolment for this study;
* Rigid or soft contact lens wearer, including orthokeratology in the last 30 days;
* Previous corneal refractive surgery;
* Pregnancy or breastfeeding.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2018-10-19 (Actual); Study Completion 2018-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Tan-Showyin, PhD, Principal Investigator — University of New South Wales
Locations (1):
- School of Optometry and Vision Science, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No
Any data included in reports, publications or presented at meetings will be provided in the form of group responses or study identity numbers, such that the participants cannot be identified.

RESULTS

PARTICIPANT FLOW:
Groups:
- Lacritec: Combination of flaxseed oil, borage oil and fish oil omega-3 fatty acids
  Lacritec: Concentrated Omega-3 Triglycerides-fish 332 mg Equiv. Eicosapentaenoic Acid (EPA) 134 mg Equiv. Docosahexaenoic Acid (DHA) 66.8 mg Flax Seed Oil (Linseed Oil) 334 mg Equiv. Oleic acid 58.5 mg Equiv. Linoleic acid 58.5 mg Equiv. Linolenic acid 192 mg Borago officinalis seed oil fixed (Borage) 434 mg Equiv. gamma-Linolenic acid 95.5 mg
Period: Overall Study
Arm/Group | Lacritec | Placebo
Started | 61 | 58
Completed | 49 | 52
Not Completed | 12 | 6

BASELINE CHARACTERISTICS:
Groups:
- Supplement: Combination of flaxseed oil, borage oil and fish oil omega-3 fatty acids
  Lacritec: Concentrated Omega-3 Triglycerides-fish 332 mg Equiv. Eicosapentaenoic Acid (EPA) 134 mg Equiv. Docosahexaenoic Acid (DHA) 66.8 mg Flax Seed Oil (Linseed Oil) 334 mg Equiv. Oleic acid 58.5 mg Equiv. Linoleic acid 58.5 mg Equiv. Linolenic acid 192 mg Borago officinalis seed oil fixed (Borage) 434 mg Equiv. gamma-Linolenic acid 95.5 mg
- Total: Total of all reporting groups
Arm/Group | Supplement | Placebo | Total
Number analyzed (Participants) | 61 | 58 | 119
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 2 | 4
  Between 18 and 65 years | 49 | 42 | 91
  >=65 years | 10 | 14 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.9 (18.2) | 44.1 (19.2) | 41.43 (18.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 37 | 81
  Male | 17 | 21 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 61 | 58 | 119
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 35 | 25 | 60
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 26 | 33 | 59
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 61 | 58 | 119
Ocular Surface Disease Index [Mean (Full Range); unit: units on a scale] — Ocular Surface Disease Index score ranges from 5 to 100. Lower scores indicates better subjective symptoms (better outcomes).
  units on a scale | 37 [21.6 to 52.4] | 36 [20.4 to 51.6] | 36 [20.4 to 52.4]
Ocular Comfort Index [Mean (Inter-Quartile Range); unit: units on a scale] — Ocular Comfort Index score ranges from 0 to 100. Lower scores indicates better subjective symptoms (better outcomes).
  units on a scale | 40.6 [25.20 to 47.6] | 38.9 [32.50 to 45.30] | 39.0 [30.35 to 47.65]
Dry Eye Questionnaire - 5 [Mean (Inter-Quartile Range); unit: units on a scale] — Dry Eye Questionnaire score ranges from 0 to 100. Lower scores indicates better subjective symptoms (better outcomes).
  units on a scale | 12.43 [9.33 to 15.53] | 11.5 [8.3 to 14.70] | 11.80 [8.45 to 15.15]
Non-invasive tear break-up time [Mean (Standard Deviation); unit: seconds] | 11.7 (5.1) | 12.0 (6.4) | 11.70 (6.28)
Tear Evaporation [Mean (Inter-Quartile Range); unit: g.m^2.h] — Tear evaporation rate ranges from 20 to 200. Lower scores indicates better subjective symptoms (better outcomes).
  g.m^2.h | 58.03 [32.17 to 83.89] | 58.36 [32.48 to 84.24] | 58.24 [33.64 to 82.80]

OUTCOME MEASURES:

1. Primary Outcome: Subjective Ocular Symptoms
Description: Measured using the Ocular Surface Disease Index questionnaire. Ocular surface disease index is assessed on a scale of 0 to 100 with higher score representing greater disability. Scores can range from 10 to 100.
Time Frame: 3 months
Population: All participant received at-least one dose of treatment.
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Lacritec | Placebo
Number analyzed (Participants) | 61 | 58
score on a scale | 27.42 [11.18 to 43.66] | 27.43 [11.8 to 43.48]

2. Primary Outcome: Subjective Ocular Comfort
Description: Measured using the Ocular Comfort Index questionnaire. Ocular comfort index questionnaire score range from 0 to 72. Lowest slow indicates better subjective symptoms.
Time Frame: 3 months
Population: All participants received at least one dose of treatment.
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Lacritec | Placebo
Number analyzed (Participants) | 61 | 58
score on a scale | 35.61 [27.08 to 44.14] | 35.66 [27.11 to 44.21]

3. Primary Outcome: Subjective Ocular Dryness
Description: Measured using the Dry Eye Questionnaire 5. Dry eye questionnaire 5 score ranges from 0 to 22.
  Lower score represents better outcome.
Time Frame: 3 months
Population: All participants received at least one dose of treatment.
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Lacritec | Placebo
Number analyzed (Participants) | 61 | 58
score on a scale | 9.75 [5.81 to 13.69] | 9.78 [5.89 to 13.67]

4. Secondary Outcome: Non-invasive Tear Film Break-up Time
Description: Measured in seconds using the Oculus Keratograph. Higher value represents better outcome.
Time Frame: 3 months
Population: All participants received at least one dose of treatment.
Measure: Mean (Inter-Quartile Range); unit: Seconds
Arm/Group | Lacritec | Placebo
Number analyzed (Participants) | 61 | 58
Seconds | 11.50 [5.84 to 17.16] | 11.49 [5.88 to 17.1]

5. Secondary Outcome: Tear Evaporation Rate
Description: Measured in g.m^2.h using the Vapometer
Time Frame: 3 months
Population: All participants received at least one dose of treatment.
Measure: Mean (Standard Deviation); unit: g.m^2.h
Arm/Group | Lacritec | Placebo
Number analyzed (Participants) | 61 | 58
g.m^2.h | 59.10 (25.41) | 59.11 (25.48)

6. Secondary Outcome: Tear Meniscus Height
Description: Measured in millimeters using the Oculus Keratograph 5M
Time Frame: 3 months
Population: All participants received at least one dose of treatment.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Lacritec | Placebo
Number analyzed (Participants) | 61 | 58
mm | 0.26 (0.10) | 0.27 (0.19)

7. Secondary Outcome: Tear Volume
Description: Measured in millimeters using phenol red thread tests
Time Frame: 3 months
Population: All participants received at least one dose of treatment.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Lacritec | Placebo
Number analyzed (Participants) | 61 | 58
mm | 18.17 (6.73) | 18.13 (6.89)

8. Secondary Outcome: Tear Film Lipid Layer Thickness
Description: Measured in nanometers using the LipiView ocular surface interferometer
Time Frame: 3 months
Population: All participants received at least one dose of treatment.
Measure: Mean (Standard Deviation); unit: nm
Arm/Group | Lacritec | Placebo
Number analyzed (Participants) | 61 | 58
nm | 64.59 (20.33) | 64.84 (19.98)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Lacritec | Placebo
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/58
Other Adverse Events (participants affected / at risk) | 13/61 | 15/58
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacritec (N=61) | Placebo (N=58)
Digestive issues (Gastrointestinal disorders) | 13 (13) | 15 (15)

LIMITATIONS AND CAVEATS:
To manufacture the placebo soft gel capsule, inclusion of oleic acid in the formulation was required, which could have an influence on the placebo arm of the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-24): https://cdn.clinicaltrials.gov/large-docs/31/NCT03141931/Prot_SAP_000.pdf